CLINICAL TRIAL: NCT01355042
Title: DYNAMICS: DNA as a Prognostic Marker in ICU Patients Study
Brief Title: Studies of Blood DNA in Patients With Severe Infection DYNAMICS
Acronym: DYNAMICS
Status: Completed | Type: Observational
Sponsor: Alison Fox-Robichaud (Other)
Responsible Party: Sponsor-Investigator, Alison Fox-Robichaud, Physician, Hamilton Health Sciences Corporation
Organization: Hamilton Health Sciences Corporation (Other)
Other Study IDs: CIHR-220268
Record Dates: First submitted 2011-05-16; First posted 2011-05-17 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Sepsis; Shock; Trauma
MeSH Terms: conditions — Sepsis; Shock; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Severe Sepsis and Septic Shock
- Other Critical Ill with or without Shock: Severe Trauma, Neurological Injury, Other Shock (not Septic)

SUMMARY:
Severe sepsis (ie. life-threatening infections) is triggered by harmful microorganisms or their toxins in the blood or tissues. These harmful agents damage the lining of blood vessels which can lead to inflammation, blood clot formation, and vessel obstruction. In Canada, there are approximately 90,000 patients with severe sepsis each year. Of these, 30% to 50% will die. The identification of highly reliable outcome predictors in severe sepsis patients is important for several reasons including: to help describe the severity of sepsis, to classify patients for enrollment in clinical studies, and to monitor a patient's response to treatment and procedures. In the investigators lab, the investigators examined the incremental usefulness of adding multiple biomarkers to clinical scoring systems for predicting ICU mortality in patients with severe sepsis. In a preliminary study of 80 patients with sepsis, the investigators found that high levels of plasma DNA predicted ICU death better than any other clinical or biological factor. In this grant, the investigators propose to confirm these findings in an external group of 400 patients in a blinded fashion. The investigators also plan to study how plasma DNA levels change over time and whether high plasma DNA levels can be used to distinguish sepsis from other critically ill conditions. For this the investigators will compare the investigators septic patients to a cohort of 600 patients in the ICU with other conditions. The investigators believe this research has the potential to significantly improve the management and treatment of septic patients.

DETAILED DESCRIPTION:
DYNAMICS STUDY (DNA as prognostic marker in ICU patients)

Principal Investigator: Patricia Liaw, PhD (McMaster University) Coinvestigator: Alison Fox-Robichaud, MD (McMaster University) Funding source: CIHR, 2010-2015 Budget: $794,086

One-page Protocol summary This is a new 5-year CIHR funded multi-centre prospective observational study. The overall objective is to gain insight into the pathophysiology of plasma DNA (ie. cell-free DNA) in severe sepsis patients and in other critically ill patients. In our pilot study of 80 severe sepsis patients, we found that plasma DNA had extremely high prognostic utility in this patient population. Using Receiver Operating Characteristic (ROC) curves in a multivariate logistic model, we demonstrated that the Area Under the Curve (AUC) for plasma DNA is 0.96 (95% CI 0.93-1.00). Furthermore, plasma DNA levels obtained at "day 1" (ie. within 24 hours of meeting the inclusion criteria for severe sepsis) did not differ significantly from the levels measured in subsequent days. In other words, plasma DNA levels in nonsurvivors were high at "day 1" and remained high; plasma DNA levels in survivors were low at "day 1" and remained low. These finding suggests that at study inclusion for severe sepsis, the nonsurvivor patients had already reached "a point of no return" (with the standard of care available at the time the patients in the pilot study were recruited).

We plan to validate the prognostic utility of plasma DNA prospectively in an independent cohort of severe sepsis patients (n=400). We will also study a broad cohort of non-septic ICU patients (n=600) to determine if elevations in plasma DNA are specific to severe sepsis, or if it is more generally associated with high mortality risk. These non-septic ICU patients include the following: multiple trauma, shock on presentation, neurosurgery, aneurysm, intracranial hemorrhage, burns). The overall research coordinator for this study is Ellen McDonald. Participating centres include Hamilton (Patricia Liaw, Alison Fox-Robichaud, Deborah Cook), Ottawa (Laurlyn McIntyre), London (Claudio Martin, Doug Fraser), Vancouver (Peter Dodek), Toronto (John Marshall, Jennifer Tsang), Laval Quebec (Francois Lallouche), and Calgary (Brent Winston).

Clinical data will be collected daily during the first week, then once a week thereafter for the duration of the patients' stay in the ICU. Blood sample will also be collected on the same schedule except that weekend blood samples will be skipped. Freezerworks Unlimited will be used for barcoding and tracking of all plasma samples. All samples will be shipped to Hamilton for biomarker analyses. Clinical data will be managed with the iDataFax software with statistical support from Janice Pogue at the Population Health and Research Institute (Hamilton). The primary outcome is ICU mortality. The secondary outcomes are (a) the temporal relationships between plasma DNA levels and other markers of inflammation and blood clotting, and (b) the temporal relationships between plasma DNA levels and clinical parameters (e.g. SOFA and MODS scores, interventions, use of blood products and plasma expanders).

This study was approved by the Research Ethics Board at the Hamilton Health Sciences in November 2010. Deferred consent has been approved. Although we are not performing any DNA sequencing analyses on the patient samples (ie. we are simply quantifying how much DNA is in the plasma), we are also collecting Paxgene DNA tubes in the event that future as-yet-undetermined studies require DNA for gene sequencing studies. Our local Ethics Board has approved a separate Genetic Consent form to request and extra blood samples for Paxgene DNA tubes. As of May 2012 we have completed recruitment in the sepsis arm. We are starting to close some sites to enrolment as we near study completion

ELIGIBILITY:
Inclusion Criteria:

* admitted to an intensive care unit with either sepsis or other critical illness in previous 24 hrs

Exclusion Criteria:

* less than 18 yrs old
* not expected to survive 72 hrs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to academic intensive care units
Sampling Method: Probability Sample
Enrollment: 792 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2012-06 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Liaw, PhD, Principal Investigator — Thrombosis and Atherosclerosis Research Institute
Locations (6):
- Canada (6):
  - Alberta Health Services -- Foothills Hospital, Calgary, Alberta
  - St. Paul's Hospital, Vancouver, British Columbia
  - Hamilton Health Sciences: General Site, Hamilton, Ontario
  - St Joseph's Health Care, Hamilton, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Centre Hospitalier de l'Universite Laval, Laval, Quebec

REFERENCES:
- [Derived] Jackson Chornenki NL, Coke R, Kwong AC, Dwivedi DJ, Xu MK, McDonald E, Marshall JC, Fox-Robichaud AE, Charbonney E, Liaw PC. Comparison of the source and prognostic utility of cfDNA in trauma and sepsis. Intensive Care Med Exp. 2019 May 22;7(1):29. doi: 10.1186/s40635-019-0251-4. PMID 31119471
- [Derived] Grin PM, Dwivedi DJ, Chathely KM, Trigatti BL, Prat A, Seidah NG, Liaw PC, Fox-Robichaud AE. Low-density lipoprotein (LDL)-dependent uptake of Gram-positive lipoteichoic acid and Gram-negative lipopolysaccharide occurs through LDL receptor. Sci Rep. 2018 Jul 12;8(1):10496. doi: 10.1038/s41598-018-28777-0. PMID 30002483